CLINICAL TRIAL: NCT05348343
Title: A Pilot Clinical 'Proof of Concept' Study of Activated Platelet-rich Plasma (PRP) in Subjects With Androgenetic Alopecia (AGA)
Brief Title: Activated PRP for Treatment of Androgenetic Alopecia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santiste Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM-001
Record Dates: First submitted 2022-04-14; First posted 2022-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Androgenetic Alopecia
Keywords: Alopecia; Hair loss; Skin
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autocontrolled Arm (Other): The subject will be treated with both the experimental treatment and the active comparator.
  Interventions: Biological: Autologous platelet-rich plasma

INTERVENTIONS:
Biological: Autologous platelet-rich plasma — PRP created using a commercially available system will be used for treatment. PEFA-PRP will be created by subjecting PRP to a pulsed electrical field in a specially designed instrument developed by sponsor. Two 9 cm2 contralateral regions of interest (ROI) on the scalp will be treated with approximately 6mL of either PRP or PEFA-PRP by subcutaneous injection.

SUMMARY:
A clinical trial to assess the effects and safety of PRP activated with pulsed electrical fields (PEFA-PRP) compared with unactivated PRP when used to treat AGA.

The design of this small-scale, phase 1b/2a clinical trial is to demonstrate that pulsed electric field activation of autologous PRP results in a controlled release of platelet growth factors and other biologically active molecules that will have a benefit effect on the non-cycling hair follicles in the treated scalp compared to non-activated PRP. This single-center, auto-controlled study will compare the clinical benefit of PEFA-PRP versus non-activated PRP treatment of male patients with AGA.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 30 and 60 years of age, inclusive
2. A clinical diagnosis of AGA (stage II to V, according to the Hamilton-Norwood Scale)
3. Non-smokers in good general health, as determined by the Investigator
4. Willing and able to tolerate multiple injections and attend all study visits
5. Willing to maintain the same hair style as at the Screening Visit for the duration of the study
6. Willing to have blood drawn.

Exclusion Criteria:

1. Clinical diagnosis of alopecia areata or other non-AGA forms of alopecia
2. Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
3. Current significant skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis) that might interfere with the study conduct or evaluations
4. History of surgical correction for hair loss such as transplantation
5. Previous exposure to Platelet-rich Plasma (PRP) for alopecia
6. Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within 30 days prior to the Screening Visit
7. Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, cimetidine) within 30 days prior to the Screening Visit
8. No history of burning, flaking, itching, and stinging of the scalp
9. History of malignancy (except basal cell and squamous cell skin cancers) or undergoing chemotherapy or radiation treatments
10. A known history of autoimmune thyroid disease, any other thyroid disorder or other autoimmune disorders that in the opinion of the investigator may interfere with the study treatment
11. Significant tendency to develop keloids or hypertrophic scarring
12. A known history of significant physical or mental disease that the Investigator feels may impact the subject's participation
13. The use of aspirin or other NSAIDs (Nonsteroidal anti-inflammatory drugs) such as Nurofen, Voltaren, Diclofenac or Naproxen 7 days before beginning each of the treatments during the study
14. The use of Vitamin E supplements (other than in multivitamins) 14 days before beginning each of the treatments during the study
15. Current anticoagulant therapy (heparins; factor Xa inhibitors; direct agents such dabigatran, rivaroxaban, apixaban, edoxaban and betrixaban; warfarin/coumarins
16. Hereditary or acquired hematological/coagulation disorders such as: platelet dysfunction syndrome, critical thrombocytopenia, hypofibrinogenemia, impaired coagulation, drepanocytosis (sickle cell anemia)
17. Utilization of low-level lasers to scalp within 90 days prior to the Screening Visit
18. Platelet count of less than 150,000 platelets/µL as measured by automated complete blood cell count and differential at or around the time of treatment (within 3 days of injection)
19. Treatment with another investigational drug or other intervention within the previous 180 days
20. Current smoker or tobacco use within the previous 2 years

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in hair density and hair regrowth | Month 6 and Month 8
  The change in hair density (hair count and thickness) measured in the region of interest (ROI) at six months and eight months using automated image analysis with Trichovision/Fotofinder imaging software. The change will be compared to the following:
  1. Baseline in the same ROI
  2. An entire treatment area with diagnosed AGA on the scalp
  3. The same region on the contralateral scalp
Measurement of hair regrowth | Month 6 and Month 8
  The amount of hair regrowth measured in the region of interest (ROI) at six months and eight months using automated image analysis with Trichovision/Fotofinder imaging software. The change will be compared to the following:
  1. Baseline in the same ROI
  2. An entire treatment area with diagnosed AGA on the scalp
  3. The same region on the contralateral scalp

SECONDARY OUTCOMES:
Clinical progression of treatment as determined by principal investigator | Month 6 and Month 8
  Global photography evaluation by the PI using Norwood Hamilton scale.
Clinical progression of treatment as determined by subject | Month 6 and Month 8
  Change in reported patient satisfaction outcome surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Maryanne M. Senna, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No